CLINICAL TRIAL: NCT07245654
Title: Monitoring the Depth of Anesthesia and Nociception During the Induction of General Anesthesia in Pediatric Patients: a Prospective Observational Study
Brief Title: Monitoring the Depth of Anesthesia and Nociception During the Induction of General Anesthesia in Pediatric Patients
Acronym: ANIGAPP
Status: Recruiting | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, prof. MUDr. Petr Štourač, Ph.D., LL.M, MBA, FESAIC, Brno University Hospital
Other Study IDs: KDAR 2025 ANIGAPP
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Anaesthesia; Anesthesia Depth Monitoring
Keywords: depth of anesthesia; pediatric; nociception; awareness; depth of analgesia; airway management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Perioperative assessment of adequate depth of anesthesia and analgesia is currently a recommended part of routine anesthesia practice for all surgical procedures. In most cases, it is performed by monitoring and evaluating physiological parameters, which is insufficient, especially for the depth of anesthesia. The depth of anesthesia, when measured with the Conox device, is indicated by the qCON index, the recommended value for anesthesia management is between 40-60. Shallow (above 60) anesthesia may be associated with an increased incidence of perioperative wakefulness episodes, and deeper (below 40) anesthesia may lead to a more frequent occurrence of adverse effects of anesthesia, including emergent delirium in the postoperative period. In addition to assessing the depth of anesthesia, the Conox device also allows for instrumental assessment of analgesia. Inadequate analgesia increases postoperative discomfort and may contribute to an increased incidence of complications in anesthesia and during the postoperative period. Instrumental monitoring of the depth of anesthesia and analgesia increases the safety of anesthesia care. During perioperative care, periods with significant painful stimulation include not only the surgical procedure itself but also airway management during induction of general anesthesia, especially intubation. The hypothesis is - due to the significant painful stimulation during airway management during induction of anesthesia, adequate depth of anesthesia and analgesia may be insufficient and is associated with the patient's clinical response, which may be associated with the occurrence of postoperative delirium.

DETAILED DESCRIPTION:
After approval by the Ethics Committee of the Brno University Hospital and registration at clinicaltrials.gov, the study will include patients meeting inclusive criteria. Pediatric patients aged 1 year to 19 years who undergo elective surgery under general anesthesia will be included in the study if the expected duration of the operation is more than 30 minutes.

Due to the observational nature of the study (no intervention, the monitoring used is a standard recommended part of anesthesia care), informed consent will not be required. Before induction of anesthesia, the electrodes of the CONOX device will be applied to the patient's forehead according to the manufacturer's recommendations and monitoring of the depth of anesthesia and analgesia will be initiated. Induction of anesthesia will be carried out according to the indications of the anesthesiologist (intravenously or by inhalation). During airway management, the depth of anesthesia and the level of analgesia and the patient's clinical response will be monitored. At the same time, the opioid analgesic used, the method of airway management and the occurrence of a burst suppression ratio will be monitored. Postoperatively, the occurrence of postoperative delirium in the recovery room will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (age 1-19 years) indicated for surgery under general anesthesia with airway management (laryngeal mask, orotracheal intubation, nasotracheal intubation)
* CONOX monitoring available

Exclusion Criteria:

* Age out of range
* Use of ketamine during anesthesia care (premedication, analgesic, anesthetic)
* Expected duration of surgery less than 30 minutes
* CONOX monitoring unavailable

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - Pediatric patients (age 1-19 years) indicated for surgery under general anesthesia with airway management (laryngeal mask, orotracheal intubation, nasotracheal intubation) with expected duration of surgery more than 30 minutes
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Depth of anesthesia | Perioperative/Periprocedural
  Assessment of the depth of anesthesia, level of analgesia during airway management during induction of anesthesia, clinical response of the patient.

SECONDARY OUTCOMES:
contributing factors | Perioperative/Periprocedural
  Evaluation of the opioid analgesic used, method of airway management, the occurrence of BSR value above 0, the occurrence of postoperative delirium during recovery from anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, prof.MD.Ph.D, Principal Investigator — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No